CLINICAL TRIAL: NCT06275399
Title: Comprehensive Assessment of Morphometric, Functional, Biomechanical, and Biological Interactions Between Atherosclerotic Plaque and Blood Platelets Within the Stenosed Coronary Artery in Vivo: a Prospective Study
Brief Title: Comprehensive Assessment of Morphometric, Functional, Biomechanical and Biological Interactions Between Atherosclerotic Plaque and Platelets Within the Stenosed Coronary Artery
Acronym: INTERFORCE
Status: Recruiting | Type: Observational
Sponsor: Medical University of Warsaw (Other)
Collaborators: National Science Centre, Poland (Other Government); University College, London (Other); Queen Mary University of London (Other)
Responsible Party: Principal Investigator, Mariusz Tomaniak, Tomaniak Mariusz MD PhD Assoc. Prof., Medical University of Warsaw
Other Study IDs: INTERFORCE
Record Dates: First submitted 2024-02-07; First posted 2024-02-23 (Actual); Last update posted 2024-02-23 (Actual); Status verified 2024-02

CONDITIONS: Chronic Coronary Syndrome; Atherosclerosis
Keywords: Optical Coherence Tomography; vFFR; Shear Rate; Impedance aggregometry; Shear stress; Proteomic; Metabolomic; Computational fluid dynamics; Prothrombotic platelet; Vulnerable plaque
MeSH Terms: conditions — Atherosclerosis | interventions — Blood Specimen Collection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Patients with chronic coronary syndrome and coronary stenosis (30% - 90%) amenable to OCT imaging: Patients with chronic coronary syndrome and coronary stenosis (30% - 90%) amenable to OCT imaging. The groups will be assessed at the time of angiography with:
  * OCT for evaluation of plaque morphology within the coronary stenosis
  * Computational fluid dynamics with vFFR and estimation of value and distribution of shear rate and shear stress
  * Impedance aggregometry based platelet reactivity
  * Single-particle high-resolution flow cytometry analysis of pMVs and sEVs as well as additional platelet activation and inflammatory biomarkers
  * Proteomic and metabolomic characterization - in the subset of patients
  Biomarker assessment will be done in the blood sampled directly from coronary artery (proximal and distal segment) arteries. Shear rate/shear stress distribution and biomarkers profile will be compared between the stenotic vessel and the non-stenotic vessel (stenoses <30%) in the same patient.
  Interventions: Diagnostic Test: OCT examination; Diagnostic Test: Blood sampling; Diagnostic Test: Assessment of vFFR and shear stress parameters

INTERVENTIONS:
Diagnostic Test: OCT examination — OCT examination for precise evaluation of plaque morphology within the coronary stenosis.
Diagnostic Test: Blood sampling — Blood sampling directly from coronary artery (proximal and distal segment) arteries
Diagnostic Test: Assessment of vFFR and shear stress parameters — The procedure is based on non-invasive assessment of vFFR and shear stress parameters with dedicated software, deriving parameters directly from coronary angiography with the calculation based on the computational fluid dynamics

SUMMARY:
The main objective of the present study is to verify, in vivo, whether shear forces computed solely based on coronary angiography and computational fluid dynamics (CFD) techniques are associated with the biomarkers indicating the prothrombotic tendency of circulating blood in situ - distally and proximally to the coronary stenosis. The study will prospectively assess the relationship between i) the value and distribution of shear rate and shear stress (SS) estimated using three-dimensional angiography and CFD techniques, and ii) atherosclerotic plaque characteristics as assessed by optical coherence tomography (OCT), iii) functional parameters of diseased vessels assessed by vessel fractional flow reserve (vFFR), and iv) in situ platelet activation, as expressed by platelet-derived microvesicles (pMVs) and small extracellular vesicles (sEVs), platelet aggregometry and other serum prothrombotic or inflammatory biomarkers sampled within the coronary artery.

DETAILED DESCRIPTION:
The biomechanical forces, including shear rate and shear stress exerted by circulating blood on the coronary wall and on circulating blood elements have been reported to contribute to the processes of plaque destabilization and thrombosis. Reliable estimation of shear (shear rate and shear stress) acting in vivo within the coronary artery has now become possible using imaging data and computational fluid dynamics techniques. The changing microenvironment of the plaque has a crucial role in the biochemical processes involved in remodeling the plaque itself. In this prospective, single-center study a total of 105 patients will be enrolled presenting with chronic coronary syndrome and angiographically confirmed coronary stenosis (30% - 90%) amenable to OCT imaging (according to the operator's judgment).

The groups will be assessed at the time of angiography with:

* OCT examination for precise evaluation of plaque morphology within the coronary stenosis
* Computational fluid dynamics with vFFR and estimation of value and distribution of shear rate and shear stress
* Impedance aggregometry-based platelet reactivity
* Single-particle high-resolution flow cytometry analysis of platelet-derived microvesicles and small extracellular vesicles (sEVs) as well as additional platelet activation (P-selectin, annexin-V) and inflammatory biomarkers
* Proteomic and metabolomic characterization - in the subset of patients Biomarker assessment will be done in the blood sampled directly from coronary artery (proximal and distal segment).

ELIGIBILITY:
Inclusion Criteria:

* Chronic coronary syndrome
* Angiographically confirmed coronary stenosis (30% - 90%)
* Amenable to OCT imaging

Exclusion Criteria:

* Cardiogenic shock
* ST-segment elevation or non-ST-segment elevation myocardial infarction
* Active bleeding
* Left main coronary artery disease
* Multivessel disease
* Lesions located at a distance ≤3 mm from the ostium of the vessel
* Thrombocytopenia
* Previous coronary artery bypass grafting
* Previous coronary intervention with stent implantation or balloon angioplasty
* Previous use of novel oral anticoagulants or vitamin K antagonists

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients will be enrolled presenting with chronic coronary syndrome and angiographically confirmed coronary stenosis (30% - 90%) amenable to OCT imaging (according to the operator's judgment).
Sampling Method: Probability Sample
Enrollment: 105 (Estimated)
Dates: Start 2023-07-21 (Actual); Primary Completion 2025-07-21 (Estimated); Study Completion 2026-07-21 (Estimated)

PRIMARY OUTCOMES:
Correlation between the mean shear rate and shear stress values at the lesion's site and the concentration of pMVs and sEVs sampled in the distal segment of the artery. | Baseline

SECONDARY OUTCOMES:
Correlation between the shear stress measurements at the site of the lesion and the concentration of inflammatory biomarkers in the distal segment of the artery | Baseline
  Inflammatory biomarkers will include sST2, sRAGE, sCD40L, sFlt-1, LIGHT, TNF-α, PlGF, IL-6, IL-18, IL-10, CCL2
Correlation between the shear stress measurements at the site of the lesion and the platelet reactivity parameters in the distal segment of the artery | Baseline
  Platelet reactivity will be defined as the area under the curve of aggregation units (AU) over time using impedance aggregometry with ADP, ASPI, and TRAP-6 tests
Correlation between the shear rate and shear stress values at the site of the lesion and the gradient (delta) concentration of the pMVs and sEVs | Baseline
Correlation between the shear rate and shear stress values at the site of the lesion and the gradient (delta) concentration of inflammatory biomarkers | Baseline
  Inflammatory biomarkers will include: sST2, sRAGE, sCD40L, sFlt-1, LIGHT, TNF-α, PlGF, IL-6, IL-18, IL-10, CCL2
Correlation between the shear rate and shear stress values at the site of the lesion and the gradient (delta) of platelet reactivity | Baseline
  Platelet reactivity will be defined as the area under the curve of aggregation units (AU) over time using impedance aggregometry with ADP, ASPI, and TRAP-6 tests
Concentrations of inflammatory biomarkers categorized by the atherosclerotic plaque morphology and the mean value of shear stress affecting the endothelium at the stenosis site and as well as according to the vessel | Baseline
  Inflammatory biomarkers will include: sST2, sRAGE, sCD40L, sFlt-1, LIGHT, TNF-α, PlGF, IL-6, IL-18, IL-10, CCL2
Platelet reactivity levels categorized by the atherosclerotic plaque morphology and the mean value of shear stress affecting the endothelium at the stenosis site and as well as according to the vessel | Baseline
  Platelet reactivity will be defined as the area under the curve of aggregation units (AU) over time using impedance aggregometry with ADP, ASPI, and TRAP-6 tests
Concentrations of pMVs and sEVs categorized by the atherosclerotic plaque morphology and the mean value of shear stress affecting the endothelium at the stenosis site and as well as according to the vessel | Baseline
Platelet reactivity levels in blood sampled from the stenosed vs. the non-stenosed coronary artery | Baseline
  Platelet reactivity will be defined as the area under the curve of aggregation units (AU) over time using impedance aggregometry with ADP, ASPI, and TRAP-6 tests
Concentrations of analyzed pMVs and sEVs in blood sampled from the stenosed vs. the non-stenosed coronary artery | Baseline
Concentrations of analyzed inflammatory biomarkers in blood sampled from the stenosed vs. the non-stenosed coronary artery | Baseline
  Inflammatory biomarkers will include: sST2, sRAGE, sCD40L, sFlt-1, LIGHT, TNF-α, PlGF, IL-6, IL-18, IL-10, CCL2
Correlation between vFFR delta pressure and the delta platelet reactivity in stenosed artery compared to these gradients in a non-stenosed artery in the same patient | Baseline
  Platelet reactivity will be defined as the area under the curve of aggregation units (AU) over time using impedance aggregometry with ADP, ASPI, and TRAP-6 tests
Correlation between vFFR delta pressure and the delta concentration of the pMVs and sEVs in stenosed artery compared to these gradients in a non-stenosed artery in the same patient | Baseline
Correlation between vFFR delta pressure and the delta concentration of the inflammatory biomarkers in stenosed artery compared to these gradients in a non-stenosed artery in the same patient | Baseline
  Inflammatory biomarkers will include: sST2, sRAGE, sCD40L, sFlt-1, LIGHT, TNF-α, PlGF, IL-6, IL-18, IL-10, CCL2

CONTACTS AND LOCATIONS:
Locations (1):
- Medical University of Warsaw, Warsaw, Masovian Voivodeship, Poland

IPD SHARING:
Plan to Share IPD: No